CLINICAL TRIAL: NCT02655614
Title: A Phase I, Double-Blind, Randomized, Placebo-Controlled, Multicenter, Single- and Multiple-Ascending-Dose Study to Determine Initial Safety, Tolerability, and Pharmacokinetics of GDC-0134 in Patients With Amyotrophic Lateral Sclerosis
Brief Title: A Study of GDC-0134 to Determine Initial Safety, Tolerability, and Pharmacokinetic Parameters in Participants With Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GN29823; 2017-002931-41 (EudraCT Number)
Record Dates: First submitted 2016-01-07; First posted 2016-01-14 (Estimated); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Rabeprazole; Midazolam; Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes

ARMS (5):
- SAD Stage: GDC-0134 (Experimental): Participants in multiple cohorts and treatment periods will receive single doses of GDC-0134 oral capsules under fed/fasting conditions. To study the effect of proton pump inhibitor (PPI) medication rabeprazole on PK properties of GDC-0134, few participants may receive rabeprazole 20 milligrams (mg).
  Interventions: Drug: GDC-0134; Drug: Rabeprazole
- SAD Stage: Placebo (Placebo Comparator): Participants in multiple cohorts and treatment periods will receive placebo matching to GDC-0134 under fed/fasting conditions. Few participants may receive rabeprazole 20 mg.
  Interventions: Drug: Placebo; Drug: Rabeprazole
- MAD Stage: GDC-0134 (Experimental): Participants will receive multiple doses of GDC-0134 for 28 days. To study the interactions between GDC-0134 and other drugs, some participants may receive single doses of midazolam and caffeine at various time points.
  Interventions: Drug: GDC-0134; Drug: Midazolam; Drug: Caffeine
- MAD Stage: Placebo (Placebo Comparator): Participants will receive placebo matching to GDC-0134 for 28 days. To study the interactions between GDC-0134 and other drugs, some participants may receive single doses of midazolam and caffeine at various time points.
  Interventions: Drug: Placebo; Drug: Midazolam; Drug: Caffeine
- Open-Label Safety Expansion (OSE) (Other): Participants will receive GDC-0134 at a dose determined by the corresponding MAD cohort.
  Interventions: Drug: GDC-0134

INTERVENTIONS:
Drug: GDC-0134 — GDC-0134 capsule will be administered orally at various doses, depending on the cohort and treatment period.
  Arms: MAD Stage: GDC-0134; Open-Label Safety Expansion (OSE); SAD Stage: GDC-0134
Drug: Placebo — Placebo matching to GDC-0134
  Arms: MAD Stage: Placebo; SAD Stage: Placebo
Drug: Rabeprazole — Rabeprazole 20 mg twice daily orally
  Arms: SAD Stage: GDC-0134; SAD Stage: Placebo
Drug: Midazolam — 2mg of liquid formulation of midazolam orally
  Arms: MAD Stage: GDC-0134; MAD Stage: Placebo
Drug: Caffeine — 100 mg tablet or solution of caffeine orally
  Arms: MAD Stage: GDC-0134; MAD Stage: Placebo

SUMMARY:
This first-in-human, double-blind, placebo-controlled Phase I study will be conducted in participants with amyotrophic lateral sclerosis (ALS) to explore safety, tolerability, and pharmacokinetic (PK) properties of GDC-0134. It will include three components: a Single-Ascending-Dose (SAD) stage, a Multiple-Ascending-Dose (MAD) stage, and an Open-Label Safety Expansion (OSE) stage.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants with a diagnosis of possible, laboratory-supported probable, probable, or definite ALS according to modified El Escorial criteria
* Upright forced vital capacity of at least 50 percent (%)
* Ability to fast from food for 8 hours prior to dosing and 2 hours after dosing

Exclusion Criteria:

* Currently taking riluzole unless on a stable dose for the 3 months prior to Day -1 and without current liver enzyme or liver function abnormalities
* Currently taking edaravone unless after completion of at least the second 14-day drug-treatment period, as long as Day 1 occurs during a drug-free period at least 24 hours after the last edaravone dose and at least 5 days prior to the first dose of the next cycle
* Positive for hepatitis C antibody, hepatitis B surface antigen, or human immunodeficiency virus (HIV) antibody
* Clinically significant thrombocytopenia
* Currently taking nutritional/herbal supplements, except for over-the-counter vitamins that are within Recommended Dietary Allowance (RDA), unless discontinued at least 7 days prior to Day -1, except upon approval of both the investigator and Sponsor
* For participants participating in a designated drug-drug interaction (DDI) cohort in the MAD stage of the study, who require midazolam/caffeine administration: known allergy, religious prohibition, or other condition limiting midazolam or caffeine administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-05-31 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) | From randomization up to approximately 48 months
Percentage of Participants With Clinically Significant Laboratory Abnormalities | From randomization up to approximately 48 months
Percentage of Participants With Clinically Significant Vital Signs Abnormalities | From randomization up to approximately 48 months
Percentage of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities | From randomization up to approximately 48 months
Percentage of Participants With Clinically Significant Abnormalities in Physical Examination Findings | From randomization up to approximately 48 months

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of GDC-0134 | From Day 1 up to 28 days after last dose
Time to Maximum Plasma Concentration (tmax) of GDC-0134 | From Day 1 up to 28 days after last dose
Area Under the Plasma Concentration Versus Time Curve (AUC) of GDC-0134 | From Day 1 up to 28 days after last dose
Apparent Clearance (CL/F) of GDC-0134 | From Day 1 up to 28 days after last dose
Apparent Terminal Volume of Distribution (Vz/F) of GDC-0134 | From Day 1 up to 28 days after last dose
Apparent Terminal Half-Life (t1/2) of GDC-0134 | From Day 1 up to 28 days after last dose
PK-Dose Proportionality of GDC-0134 as Assessed With Cmax and AUC | From Day 1 up to 28 days after last dose
Accumulation Ratio of GDC-0134 | From Day 1 up to 28 days after last dose
Dose Normalized Cmax (Cmax/Dose) of GDC-0134 | From Day 1 up to 28 days after last dose
Dose Normalized AUC (AUC/Dose) of GDC-0134 | From Day 1 up to 28 days after last dose
t1/2 of Midazolam | From Day -1 up to 28 days after last dose
t1/2 of 1-Hydroxymidazolam (Metabolite of Midazolam) | From Day -1 up to 28 days after last dose
t1/2 of Caffeine | From Day -1 up to 28 days after last dose
t1/2 of Paraxanthine (Metabolite of Caffeine) | From Day -1 up to 28 days after last dose

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (10):
- United States (8):
  - Forbes Norris Mda/als Ctr; Research Center, San Francisco, California
  - Mayo Clinic Hospital - Florida, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - The Emory ALS Clinic, Atlanta, Georgia
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Wake Research Associates, Raleigh, North Carolina
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
- MUCH - Montreal Neurological Institute & Hospital, Montreal, Quebec, Canada
- UMC Utrecht, Utrecht, Netherlands